CLINICAL TRIAL: NCT01027429
Title: Simplified Antibiotic Regimens for the Management of Sepsis in Young Infants in First-level Facilities: Randomized Controlled Trial
Brief Title: Simplified Antibiotic Therapy for Sepsis in Young Infants
Acronym: SATT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Save the Children (Other); World Health Organization (Other); London School of Hygiene and Tropical Medicine (Other); Emory University (Other)
Responsible Party: Principal Investigator, Anita Kaniz Mehdi Zaidi, Professor and Chair, Department of Paediatrics and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC134GL50124
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Neonatal Sepsis; Sepsis; Infection
Keywords: infant; newborn; sepsis; infection; community
MeSH Terms: conditions — Neonatal Sepsis; Sepsis; Infections | interventions — Penicillin G Procaine; Gentamicins; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- procaine penicillin and gentamicin (Active Comparator): Procaine penicillin, 50,000 IU/kg by intramuscular injection plus gentamicin, 5 mg/kg intramuscular injection, both given once daily for 7 days
  Interventions: Drug: procaine penicillin and gentamicin; Drug: procaine penicillin, gentamicin, amoxicillin
- Amoxicillin and gentamicin (Experimental): Oral amoxicillin (80-90 mg/kg) divided twice daily and intramuscular gentamicin, 5 mg/kg once daily, both given for 7 days
  Interventions: Drug: amoxicillin and gentamicin; Drug: procaine penicillin, gentamicin, amoxicillin
- procaine penicillin, gentamicin, and amoxicillin (Experimental): procaine penicillin, 50,000 IU/kg once daily intramuscular injection plus gentamicin 5 mg/kg once daily intramuscular injection for 2 days, followed by 5 days of oral amoxicillin, 80-90 mg/kg divided in two doses.
  Interventions: Drug: procaine penicillin, gentamicin, amoxicillin

INTERVENTIONS:
Drug: procaine penicillin and gentamicin — procaine penicillin 50,000 units/kg by intramuscular injection once daily for 7 days; gentamicin, 5 mg/kg once daily by intramuscular injection for 7 days
  Arms: procaine penicillin and gentamicin
Drug: amoxicillin and gentamicin — oral amoxicillin 80-90 mg/kg divided in two doses for 7 days intramuscular gentamicin, 5 mg/kg once daily for 7 days
  Arms: Amoxicillin and gentamicin
Drug: procaine penicillin, gentamicin, amoxicillin — procaine penicillin, 50,000 IU/kg once daily intramuscular injection plus gentamicin 5 mg/kg once daily intramuscular injection for 2 days, followed by 5 days of oral amoxicillin, 80-90 mg/kg divided in two doses.

SUMMARY:
This trial evaluates primary care clinic-based simplified antibiotic therapy options for young infants, 0-59 days old in high neonatal mortality settings in peri-urban Karachi where hospital referral is frequently refused by families.

DETAILED DESCRIPTION:
Primary Objective

To evaluate if out-patient (clinic-based) therapy of young infants with possible serious bacterial infection with 7 days of intramuscular procaine penicillin and gentamicin (reference therapy) is equivalent to:

* (1) injectable gentamicin once daily and oral amoxicillin twice daily for seven days;
* (2) injectable penicillin and gentamicin once daily for two days followed by oral amoxicillin twice daily for five days; and

Hypothesis

The proportion of babies who fail therapy at (or before 7) days will be 10% in each group. A 5% or less difference in failure rates will be considered equivalent.

Study Design

This will be a randomized, three arm, open-label equivalence trial among young infants, 0-59 days of age who are diagnosed as having possible serious bacterial infection in one of the Karachi field clinics, and whose families refuse facilitated hospital referral, and the infants meet other specified inclusion criteria.

Eligible young infants will be recruited from among those referred to the clinics by trained community health workers as having clinical signs predictive of possible serious illness during regular home visits in the surveillance area, or those presenting directly to the clinics from the areas under pregnancy and newborn surveillance. A diagnosis of possible sepsis will be made by clinicians if specified clinical criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Infants 0-59 days old who are residents of catchment population of the study hospitals or clinics
  * One or more of the following five signs: severe chest in-drawing, axillary temperature >38.0C or <35.50 C, movement only when stimulated, and history of feeding problems (confirmed by poor suck on feeding assessment)
  * Family refuses recommended hospitalization or hospitalization otherwise not feasible
  * Informed consent by a legal guardian.
* Exclusion Criteria:

Very severe infection/disease characterized by presence of any of the following signs (unconscious, convulsions, unable to feed, apnea, unable to cry, cyanosis, bulging fontanel, prolonged capillary refill, major congenital malformations, major bleeding, surgical conditions needing hospital referral, persistent vomiting defined as vomiting following three attempts to feed the baby within ½ hour)

* Very low birth weight: weight <1500
* Hospitalization for illness in the last two weeks
* Previous inclusion in the study

Max Age: 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2543 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Treatment failure | within 7 days of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Shiyam S Sunder, MBBS, Study Director — Aga Khan University
Locations (1):
- Ali Akber Shah Goth, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Longombe AL, Ayede AI, Marete I, Mir F, Ejembi CL, Shahidullah M, Adejuyigbe EA, Wammanda RD, Tshefu A, Esamai F, Zaidi AK, Baqui AH, Cousens S. Oral amoxicillin plus gentamicin regimens may be superior to the procaine-penicillin plus gentamicin regimens for treatment of young infants with possible serious bacterial infection when referral is not feasible: Pooled analysis from three trials in Africa and Asia. J Glob Health. 2022 Nov 21;12:04084. doi: 10.7189/jogh.12.04084. PMID 36403158
- [Derived] Mir F, Pearce RE, Baig-Ansari N, Qazi S, Barrett JS, Abdel-Rahman S, Kearns G, Zaidi AK. Serum amoxicillin levels in young infants (0-59 days) with sepsis treated with oral amoxicillin. Arch Dis Child. 2020 Dec;105(12):1208-1214. doi: 10.1136/archdischild-2019-317342. Epub 2020 May 13. PMID 32404437
- [Derived] Mir F, Nisar I, Tikmani SS, Baloch B, Shakoor S, Jehan F, Ahmed I, Cousens S, Zaidi AK. Simplified antibiotic regimens for treatment of clinical severe infection in the outpatient setting when referral is not possible for young infants in Pakistan (Simplified Antibiotic Therapy Trial [SATT]): a randomised, open-label, equivalence trial. Lancet Glob Health. 2017 Feb;5(2):e177-e185. doi: 10.1016/S2214-109X(16)30335-7. Epub 2016 Dec 15. PMID 27988146
- [Derived] Zaidi AK, Tikmani SS, Sultana S, Baloch B, Kazi M, Rehman H, Karimi K, Jehan F, Ahmed I, Cousens S. Simplified antibiotic regimens for the management of clinically diagnosed severe infections in newborns and young infants in first-level facilities in Karachi, Pakistan: study design for an outpatient randomized controlled equivalence trial. Pediatr Infect Dis J. 2013 Sep;32 Suppl 1(Suppl 1 Innovative Treatment Regimens for Severe Infections in Young Infants):S19-25. doi: 10.1097/INF.0b013e31829ff7aa. PMID 23945571